CLINICAL TRIAL: NCT00549900
Title: Safety and Immunogenicity Study of the HPV Vaccine (GSK-580299) in Healthy, Chinese, Female Subjects
Brief Title: A Single Centre Study to Evaluate the Safety and Immunogenicity of the Human Papillomavirus Vaccine (GSK-580299) in Chinese Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 107336
Record Dates: First submitted 2007-10-18; First posted 2007-10-26 (Estimated); Results first posted 2009-12-17 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-10

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine,; Cervical cancer; Human papillomavirus infection,
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- Cervarix Group (Experimental): Subjects received 3 doses of GSK580299 vaccine (Cervarix™, HPV -16/18 L1 VLP AS04 vaccine) according to a 0, 1, 6-month schedule.
  Interventions: Biological: GSK580299 (Cervarix™ , HPV -16/18 L1 VLP AS04 vaccine)

INTERVENTIONS:
Biological: GSK580299 (Cervarix™ , HPV -16/18 L1 VLP AS04 vaccine) — Intramuscular injection, 3 doses
  Other Names: GlaxoSmithKline Biologicals' HPV -16/18 L1 VLP AS04 vaccine

SUMMARY:
A phase I, open label, single-centre study to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' HPV -16/18 L1 VLP AS04 vaccine (GSK 580299, Cervarix TM), administered intramuscularly according to a 0, 1, 6-month schedule in healthy Chinese female subjects aged 15 - 45 years.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The rationale for the protocol posting amendment was to change the study population from 18-35 to 15-45 years and to allow subjects who were administered routine vaccines e.g. Hepatitis A&B vaccines, meningococcal vaccines, Tetanus vaccine, Diphteria Tetanus Pertussis etc. up to 8 days before each HPV dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A female of Chinese origin, residing in China, aged between 15 - 45 years (inclusive) at the time of the first vaccination.
* Written informed consent obtained from the subject. For subjects below the legal age of consent, written informed consent must be obtained from the subject's parent or Legally Acceptable Representative (LAR), and written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects must be of non-childbearing potential, or if the subject is of childbearing potential, she must be abstinent or must be using adequate contraception for 30 days prior to vaccination and continue for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days preceding and 30 days after the first dose of vaccine. Administration of some routine vaccines up to 8 days before the first dose of study vaccine is allowed.
* Previous administration of components of the investigational vaccine.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Known acute or chronic, clinically significant system conditions.
* Cancer or autoimmune disease under treatment.
* Acute disease at the time of enrolment.
* History of chronic alcohol consumption and/or drug abuse.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12-02; Primary Completion 2008-07-12 (Actual); Study Completion 2008-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Jintan, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Zhu FC, Li CG, Pan HX, Zhang YJ, Bi D, Tang HW, Datta S. Safety and immunogenicity of human papillomavirus-16/18 AS04-adjuvanted vaccine in healthy Chinese females aged 15 to 45 years: a phase I trial. Chin J Cancer. 2011 Aug;30(8):559-64. doi: 10.5732/cjc.010.10564. PMID 21801604
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107336 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix Group
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (up to Month 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Participants | 1

2. Primary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 7-day (Day 0-6) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Participants
  Pain | 26
  Redness | 16
  Swelling | 9

3. Primary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash, and urticaria.
Time Frame: During the 7-day (Day 0-6) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Participants
  Arthralgia | 2
  Fatigue | 10
  Axillary fever greater than 37 degrees Celcius | 1
  Gastrointestinal symptoms | 4
  Headache | 8
  Myalgia | 7
  Rash | 1
  Urticaria | 0

4. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is defined as any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 30 days (Day 0-29) after any vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Participants | 4

5. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Hematological Parameters
Description: Hematological and biochemical parameters assessed in blood samples include alanine aminotransferase (ALT), basophils, creatinine, eosinophils, hematocrit, lymphocytes, monocytes, neutrophils, platelets, red blood cell, and white blood cells.
  Abnormalities reported include values outside the normal ranges: values higher than normal are designated as "Above" and values lower than normal as "Below".
Time Frame: At Month 0 and Month 7
Population: Analysis was performed on subjects from the Total vaccinated cohort that completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 29
Participants
  ALT Above [Month 0] | 3
  ALT Below [Month 0] | 0
  ALT Above [Month 7] | 1
  ALT Below [Month 7] | 0
  Basophils Above [Month 0] | 0
  Basophils Below [Month 0] | 0
  Basophils Above [Month 7] | 0
  Basophils Below [Month 7] | 0
  Creatinine Above [Month 0] | 0
  Creatinine Below [Month 0] | 0
  Creatinine Above [Month 7] | 3
  Creatinine Below [Month 7] | 0
  Eosinophils Above [Month 0] | 2
  Eosinophils Below [Month 0] | 0
  Eosinophils Above [Month 7] | 0
  Eosinophils Below [Month 7] | 0
  Hematocrit Above [Month 0] | 0
  Hematocrit Below [Month 0] | 0
  Hematocrit Above [Month 7] | 0
  Hematocrit Below [Month 7] | 13
  Lymphocytes Above [Month 0] | 1
  Lymphocytes Below [Month 0] | 0
  Lymphocytes Above [Month 7] | 0
  Lymphocytes Below [Month 7] | 0
  Monocytes Above [Month 0] | 0
  Monocytes Below [Month 0] | 0
  Monocytes Above [Month 7] | 0
  Monocytes Below [Month 7] | 0
  Neutrophils Above [Month 0] | 1
  Neutrophils Below [Month 0] | 1
  Neutrophils Above [Month 7] | 2
  Neutrophils Below [Month 7] | 2
  Platelets Above [Month 0] | 3
  Platelets Below [Month 0] | 2
  Platelets Above [Month 7] | 1
  Platelets Below [Month 7] | 1
  Red blood cells Above [Month 0] | 0
  Red blood cells Below [Month 0] | 0
  Red blood cells Above [Month 7] | 0
  Red blood cells Below [Month 7] | 0
  White blood cells Above [Month 0] | 2
  White blood cells Below [Month 0] | 0
  White blood cells Above [Month 7] | 2
  White blood cells Below [Month 7] | 1

6. Primary Outcome: Number of Subjects Reporting Medically Significant Adverse Events
Description: Medically significant AEs were defined as AEs prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that were not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Throughout the study period (up to Month7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 30
Participants | 2

ADVERSE EVENTS:
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=30)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=30)
Pain (General disorders) | 26
Redness (General disorders) | 16
Swelling (General disorders) | 9
Arthralgia (General disorders) | 2
Fatigue (General disorders) | 10
Gastrointestinal symptoms (General disorders) | 4
Headache (General disorders) | 8
Myalgia (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.